CLINICAL TRIAL: NCT02240459
Title: A Double Blind, Randomized Four Way Cross Over Study to Compare the Effect of Fesoterodine 4mg and 8mg Once Daily and Oxybutynin 5mg Twice Daily After Steady State Dosing Versus Placebo on Cognitive Function in Subjects With Overactive Bladder, Over the Age of 75 Years With Mild Cognitive Impairment
Brief Title: A Study of Fesoterodine and Oxybutynin on Cognitive Function in Mild Cognitive Impairment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Adrian Wagg, Research Chair in Healthy Aging, University of Alberta
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: FES-COG 1808
Record Dates: First submitted 2014-09-11; First posted 2014-09-15 (Estimated); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Overactive Bladder; Mild Cognitive Impairment
Keywords: crossover study; placebo controlled; double blind; overactive bladder
MeSH Terms: conditions — Urinary Bladder, Overactive; Cognitive Dysfunction | interventions — fesoterodine; oxybutynin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Fesoterodine 4mg daily (Experimental): fesoterodine 4mg oral
  Interventions: Drug: fesoterodine 4mg; Drug: Oxybutynin; Drug: placebo; Drug: fesoterodine 8mg
- Fesoterodine 8mg (Experimental): Fesoterodine 8mg in form of 2, 4mg tablets
  Interventions: Drug: fesoterodine 4mg; Drug: Oxybutynin; Drug: placebo; Drug: fesoterodine 8mg
- oxybutynin (Active Comparator): oxybutynin immediate release, encapsulated 2, 5mg capsules daily
  Interventions: Drug: fesoterodine 4mg; Drug: Oxybutynin; Drug: placebo; Drug: fesoterodine 8mg
- placebo capsule (Placebo Comparator): placebo capsule, 2 per day
  Interventions: Drug: fesoterodine 4mg; Drug: Oxybutynin; Drug: placebo; Drug: fesoterodine 8mg

INTERVENTIONS:
Drug: fesoterodine 4mg — 7 days therapy followed by seven days washout. Each 4mg tablet is taken in the morning
  Other Names: Toviaz
Drug: Oxybutynin — 5mg IR oxybutynin taken bid, encapsulated into a form indistinguishable from placebo
  Other Names: ditropan
Drug: placebo — placebo capsule, one twice daily, and 2 placebo fesoterodine tablets taken each morning for masking and comparator purposes
  Other Names: placebo capsule
Drug: fesoterodine 8mg — 2, 4mg fesoterodine capsules taken together in the morning
  Other Names: Toviaz 8mg

SUMMARY:
The purpose of this study is to assess the effects of fesoterodine at 4mg and 8mg doses versus a placebo and oxybutynin 5mg bid versus placebo on cognitive abilities in older people with overactive bladder and mild cognitive impairment.

DETAILED DESCRIPTION:
This is a randomized placebo controlled, blinded four way cross over trial of the effect of medications used to treat overactive bladder on the cognition of older men and women with mild cognitive impairment. Each treatment phase is a week, with a weeks washout period before starting the next treatment. Cognitive testing is by way of a validated computer assisted battery of tests

ELIGIBILITY:
Inclusion Criteria:

1. The subject is either male or female and ≥ 75 years of age.
2. The subject has OAB as determined by ICS criteria
3. The subject has mild cognitive impairment as determined by NIA criteria
4. The subject is competent to give informed consent and perform the tasks associated with the study
5. The subject has a body mass index (BMI) between 18.0 to 30.0 kg/m2 inclusive.
6. Written informed consent has been obtained.
7. The subject is available to complete the study.
8. At training visits (visit 2): the subject has performed at or above the minimum level on at least one occasion for each individual task measure in cognitive function test training.

Exclusion Criteria:

1. The subject does not have OAB.
2. The subject has either dementia or moderate to severe cognitive impairment at screening.
3. The subject has probable clinical depression as determined by Geriatric Depression Scale (GDS) short form >5 at screening.
4. Subjects taking any cognitive enhancers (cholinesterase inhibitors or memantine).
5. The subject has a history of allergy to the study drug(s), to any component of the dosage form or any other allergy, which, in the opinion of the Investigator, contraindicates their participation.
6. The subject has any clinically significant abnormal heart rate or blood pressure measurements, at the screening visit, which, in the opinion of the Investigator, prevent safe participation in the study. (dBP< 60mmHg or > 90mmHg, sBP < 95mmHg or > 160mmHg or HR < 40bpm or > 100bpm).
7. Subjects with known history of urinary retention, severe gastrointestinal obstruction (including paralytic ileus or intestinal atony) or severe gastrointestinal conditions (including toxic megacolon or ulcerative colitis), myasthenia gravis, uncontrolled narrow angle glaucoma or shallow interior chamber or subjects deemed to be at risk for these conditions.
8. Subjects undergoing haemodialysis or who have severe renal impairment.
9. Subjects with severe hepatic impairment, defined as Child-Pugh grade IV.
10. Subjects taking potent CYP 3A4 inhibitors which would, under normal circumstances, require adjustment of the dose of the test drugs.
11. Subject has taken prescribed medication within 14 days prior to the first study day or over-the-counter medicine (including vitamins and herbal remedies) within 48 hours prior to the first study day, which in the opinion of the Investigator, will interfere with the study procedures or compromise safety.
12. Subject has an average weekly alcohol intake of greater than 21 units (male) or 14 units (female) within the 90 days prior to the study. 1 unit is 270cc of beer, 40cc of spirits or 125cc of wine.
13. History of smoking more than 10 cigarettes (or the equivalent amount of tobacco) per day within the 90 days prior to the study.
14. Subject has participated in any clinical study within the last 90 days.
15. Any clinically significant abnormality following Investigator review of the pre study physical examination.
16. Any clinical condition, which, in the opinion of the Investigator, would not allow safe completion of the study.
17. Any subjects who, in the opinion of the investigator, may find it difficult to adhere to the provisions of treatment and observation specified in the protocol.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-08; Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
continuity of attention | 1 and 4h post dose
  Continuity of Attention:
  Accuracy of responding in Choice Reaction Time task Percent Target Detection in Digit Vigilance task False Alarms in Digit Vigilance task

SECONDARY OUTCOMES:
cognitive function | 1 and 4h post last dose of study drug
  includes the following domains of cognition
  * power of attention,
  * quality of working memory,
  * quality of episodic secondary memory,
  * speed of memory
  * Montreal Cognitive assessment score

CONTACTS AND LOCATIONS:
Overall Officials: Adrian S Wagg, MD, Principal Investigator — University of Alberta
Locations (1):
- Division of Geriatric Medicine, Clinical Sciences Building, University of Alberta Hosp, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Wagg A, Dale M, Tretter R, Stow B, Compion G. Randomised, multicentre, placebo-controlled, double-blind crossover study investigating the effect of solifenacin and oxybutynin in elderly people with mild cognitive impairment: the SENIOR study. Eur Urol. 2013 Jul;64(1):74-81. doi: 10.1016/j.eururo.2013.01.002. Epub 2013 Jan 11. PMID 23332882
- [Background] Wesnes KA, Edgar C, Tretter RN, Bolodeoku J. Exploratory pilot study assessing the risk of cognitive impairment or sedation in the elderly following single doses of solifenacin 10 mg. Expert Opin Drug Saf. 2009 Nov;8(6):615-26. doi: 10.1517/14740330903260790. PMID 19747069